CLINICAL TRIAL: NCT05306431
Title: Comparison of Antimicrobial Action of Sodium Hypochlorite and Polyhexamethylene Biguanide as Root Canal Irrigants in Patients Reporting With Non-vital Necrotic Pulp and Apical Periodontitis
Brief Title: Comparison of Antimicrobial Action of Sodium Hypochlorite and Polyhexamethylene Biguanide as Root Canal Irrigants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Root canal Irrigiant
Record Dates: First submitted 2022-03-19; First posted 2022-04-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — polihexanide; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The microbiologist will be kept blind to avoid risk of bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyhexamethylene biguanide (Experimental): Polyhexamethylene biguanide (PHMB), is a disinfectant solution having a broad spectrum of antimicrobial activity and is investigated as an endodontic irrigant. It is non-corrosive, non-toxic and acts by disrupting cell membrane integrity. PHMB 0.2% has been recently used as a root canal irrigant in vitro and has shown promising results of antimicrobial effectiveness of > 99.9% for both PHMB and Sodium hypochlorite
  Interventions: Drug: Polyhexamethylene biguanide
- Sodium Hypochloride (Experimental): A number of irrigant solution has thus been proposed to serve the purpose, the most popular being sodium hypochlorite (NaOCl) because of its excellent antimicrobial activity but also the ability to dissolve organic matter.
  Interventions: Drug: Sodium Hypochlorite

INTERVENTIONS:
Drug: Polyhexamethylene biguanide — Polyhexamethylene biguanide (PHMB), is a disinfectant solution having a broad spectrum of antimicrobial activity and is investigated as an endodontic irrigant
  Other Names: PHMB
  Arms: Polyhexamethylene biguanide
Drug: Sodium Hypochlorite — A number of irrigant solution has thus been proposed to serve the purpose, the most popular being sodium hypochlorite (NaOCl) because of its excellent antimicrobial activity but also the ability to dissolve organic matter
  Other Names: Bleach
  Arms: Sodium Hypochloride

SUMMARY:
The aim of this randomized clinical trial is to compare the antibacterial effects of sodium hypochlorite (NaOCl) and Polyhexamethylene biguanide during root canal treatment .

DETAILED DESCRIPTION:
This study will compare the antibacterial effectiveness of sodium hypochlorite and PHMB, to find out whether PHMB can be used as a substitute to NaOCL. Polyhexamethylene biguanide (PHMB), is a disinfectant solution having a broad spectrum of antimicrobial activity and is investigated as an endodontic irrigant. It is non-corrosive, non-toxic and acts by disrupting cell membrane integrity.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 to 50 years

  * Both male and female patients
  * Periodontally healthy teeth as determined by Periodontal Probing
  * Patients with non-vital necrotic pulps as determined by Cold Test
  * Patients with acute apical periodontitis determined by history and clinical examination
  * Clinical Findings:

Visual: Carious tooth decay Occlusion: Hyperocclusion Pulp vitality test: Negative Periapical radiograph: Caries involving pulp space and PDL widening Percussion Test: Positive Palpation Test: Negative

• Single rooted teeth as determined radiographically

Exclusion Criteria:

* • Multirooted teeth

  * Teeth undergoing Re-endo treatments
  * Teeth with root fractures and/ non restorable determined by clinical and radiographic examination
  * Patients receiving antibiotic treatment in the past 3 months determined by history
  * Patient with Diabetes determined by history
  * Patient with history of smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Bacterial load assessed by culture | 24 hours
  Effectiveness of irrigant will be evaluated with the existence or non-existence of bacteria: Positive Effect = no bacteria exist, Negative Effect = bacteria exist. Bacterial analysis will be performed by counting the number of colonies of bacteria in the specimen: No growth = no colonies seen, Few growths = less than 10 colonies of bacteria seen, Moderate growth = less than 100 colonies more than 10 colonies of bacteria seen, Heavy growth = more than 100 colonies of bacteria seen.

CONTACTS AND LOCATIONS:
Locations (1):
- Hira Danish, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No